CLINICAL TRIAL: NCT00298714
Title: Effect of Long-Term Administration of Oral Losartan on Hepatic Fibrogenesis and Gene Expression in Chronic Hepatitis C With Significant Liver Fibrosis.
Brief Title: Effects of Losartan on Hepatic Fibrogenesis in Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARAHEPC; Protocol number: 02-0491
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Hepatitis C; Liver Fibrosis
Keywords: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — Losartan

INTERVENTIONS:
Drug: Losartan

SUMMARY:
There is evidence on the beneficial effects of the administration of angiotensin II type 1 (AT1) receptors antagonists on liver fibrosis in hepatic stellate cells, experimental models of liver fibrosis in rodents and limited information in chronic hepatitis C with mild fibrosis.

The purpose of this study is to investigate the effect of long-term administration of oral Losartan, an AT1 receptor antagonist, on liver fibrogenesis in patients with chronic hepatitis C and fibrosis F2-F3 (METAVIR score).

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 65 years
* chronic hepatitis C with intermediate fibrosis (F2-F3 in Metavir score).
* non-responder or contraindication to antiviral therapy.

Exclusion Criteria:

* any other cause of liver disease
* HIV positive
* alcohol consumption
* arterial hypertension
* creatinine > 1.5mg/dL
* treatment with AT1 receptor antagonists or angiotensin converting enzyme inhibitors in the past 12 months.
* antiviral therapy in the past 12 months
* contraindications to oral losartan

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Assessment of liver fibrogenesis by changes in gene expression of key mediators of liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, M.D., Principal Investigator — Liver Unit, Institut Clínic de Malalties Digestives, Hospital Clínic, Barcelona; Vicente Arroyo, M.D., Study Chair — Liver Unit, Institut Clínic de Malalties Digestives, Hospital Clínic, Barcelona

REFERENCES:
- [Derived] Colmenero J, Bataller R, Sancho-Bru P, Dominguez M, Moreno M, Forns X, Bruguera M, Arroyo V, Brenner DA, Gines P. Effects of losartan on hepatic expression of nonphagocytic NADPH oxidase and fibrogenic genes in patients with chronic hepatitis C. Am J Physiol Gastrointest Liver Physiol. 2009 Oct;297(4):G726-34. doi: 10.1152/ajpgi.00162.2009. Epub 2009 Jul 23. PMID 19628656